CLINICAL TRIAL: NCT03719898
Title: A Phase II Study of Brigatinib in Relapsed or Refractory ALK-Positive Anaplastic Large Cell Lymphoma
Brief Title: Brigatinib in Relapsed or Refractory ALK-Positive Anaplastic Large Cell Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-117; 18-1032 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2018-10-16; First posted 2018-10-25 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Anaplastic Large Cell Lymphoma, ALK-Positive
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic | interventions — brigatinib

STUDY DESIGN:
Intervention Model Description: Refractory or relapsed ALK positive ALCL patients who may or my not have previously received treatment with any ALK inhibitor for any indication
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Brigatinib (Experimental): 90 mg daily orally for 7 days, then 180 mg daily orally during first cycle; 180 daily orally thereafter during every subsequent cycle. Each cycle has 28 days
  Interventions: Drug: Brigatinib

INTERVENTIONS:
Drug: Brigatinib — Brigatininb is administered in tablet form. It is to be taken until disease progression, unacceptable toxicity or completion of 24 cycles. patients may continue to take brigatininb beyond 24 cycles if they are benefiting from the drug

SUMMARY:
FDA approved drugs to treat patients with relapsed or refractory anaplastic large cell lymphoma (ALCL) has a median progression free survival of 20 months. Majority of patients relapse in 2 years. This study will evaluate overall response rate of next generation ALK inhibitor brigatinib in ALK positive ALCL patients by overcoming mechanisms of resistance to ALK inhibitors on cancer patients.

DETAILED DESCRIPTION:
Although patients with ALK+ anaplastic large cell lymphoma (ALCL), a type of peripheral T-cell lymphoma (PTCL), are considered to have a favorable prognosis, relapse is not uncommon if multiple International Prognostic Index (IPI) risk factors, age ≥ 40, and beta-2 microglobulin ≥ 3 mg/L are present at diagnosis. For patients older than 40 years at diagnosis and beta-2 microglobulin ≥ 3 mg/L, progression-free survival (PFS) and overall survival (OS) is less than 50% at 2.5 years when treated with standard anthracycline-based induction therapy. Patients with ALK+ ALCL with 3 or more IPI risk factors have a 5-year PFS rate of only 20% to 30%. In total, approximately 40 to 65% of patients with ALCL develop recurrent disease after front-line chemotherapy and at relapse, the disease is historically resistant to conventional chemotherapy.

Current FDA approved for treatment of relapsed or refractory PTCLs have a median PFS of 20 months and majority of patients relapse within 2 years. Despite ALK tyrosine kinase being an attractive target for management of relapsed or refractory ALK+ ALCL, ALK gene rearrangement makes cancer resistant to first and 2nd generation ALK inhibitors. Brigatinib is a next generation inhibitor with broad activity aganst a broad spetrum of resistant ALK mutants. Brigatinib has been shown to overcome mechanisms associated with resistane to 1st and 2nd generation ALK inhibitors. It is approved as 2nd line of treament in non small cell lung cancer patients. and is being tested in patients with relapsed or refractory ALK-positive ALCL.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically confirmed diagnosis of relapsed or refractory ALCL with documented ALK+ status
2. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension in accordance with RECIL 2017 criteria as described in detail in section 11.0
3. Ongoing toxicities from prior therapy must be resolved to ≤ grade 1 (with the exceptions of grade 2 peripheral neuropathy and/or alopecia). Patients with existing toxicities that are non-significant even though greater than grade 1 can be enrolled after discussion with the sponsor-investigator.
4. Age > 18 years.
5. ECOG performance status 0-2
6. Prior use of ALK inhibitors aside from brigatinib is permitted but 8 patients enrolled need to be ALK inhibitor treatment naive
7. Patients with no archival tissue available must be agreeable to fresh biopsy at baseline.
8. Patients with a known history of HIV are permitted provided the CD4 count ≥ 100 cells/µL and serum HIV viral load < 50 copies/mL. Patients must be on stable combination antiretroviral therapy at the time of treatment initiation.
9. Patients must have normal organ and marrow function as defined below

   * Absolute neutrophil count > 1,000/mcL
   * Platelets > 75,000/mcL (or 50,000/mcL if known bone marrow involvement by lymphoma)
   * Total bilirubin within normal institutional limits (up to 2x ULN if history of Gilbert's syndrome or known liver involvement)
   * AST/ALT (SGOT/SGPT) < 2 times institutional normal limits
   * Creatinine within 1.5 x upper limit of normal institutional limits OR
   * Creatinine clearance > 30 ml/min/1.73 m2 for patients with creatinine levels above 1.5x upper institutional normal
   * Serum lipase/amylase ≤1.5 × ULN
   * Hemoglobin ≥10 g/dL (can be transfused to achieve Hgb ≥10 g/dL)
10. Ability to understand and willingness to sign a written informed consent and HIPAA consent document. LARs are allowed to sign on patient's behalf with proper documentation.
11. Female patients who are postmenopausal for at least 1 year before the screening visit, or are surgically sterile. Female patients of childbearing potential should agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse.
12. Male patients, even if surgically sterilized (i.e., status post-vasectomy), who agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug.

Exclusion Criteria:

1. History of another active primary malignancy within 2 years of initiating study treatment with the exception of non-melanomatous skin cancer, or any cancer that in the judgment of the investigator has been treated with curative intent and will not interfere with the study treatment plan and response assessment.
2. Patients who have received chemotherapy or radiation therapy within 2 weeks of initiating study treatment.
3. Patients may not be receiving any other investigational agents.
4. Patients who have symptomatic CNS metastases (parenchymal or leptomeningeal) at screening or asymptomatic disease requiring an increasing dose of corticosteroids to control symptoms within 7 days prior to randomization.

   Note: If a patient has worsening neurological symptoms or signs due to CNS metastasis, the patient needs to complete local therapy and be neurologically stable (with no requirement for an increasing dose of corticosteroids or use of anticonvulsants) for 7 days prior to enrollment.
5. History of allergic reactions attributed to other ALK inhibitors
6. History of interstitial pneumonitis or drug-related pneumonitis
7. Impaired gastrointestinal function that may affect oral absorption of brigatinib
8. Patients with known active Hepatitis B or Hepatitis C (defined as having a detectable hepatitis B or C viral load)
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Physician's discretion may be exercised to determine eligibility for patients with psychiatric illness/social situations.
10. Pregnant or breast-feeding. Refer to section 4.4 for further detail.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
objective response rate | 2 years
  proportion of patients with tumor size reduction of a predefined amount and for a minimum time period measured using RECIL 2017 criteria

SECONDARY OUTCOMES:
To assess the incidence of adverse events as assessed by NCI CTCAE v5.0 for 2 years | 2 years
  Adverse events will be documented by NCI CTCAE v 5.0 criteria
To measure the overall survival (OS) at 1 and 2 years from treatment initiation | 5 years
  Overall survival will be measured as the length of time patients survive from the day of treatment.
To measure progression-free survival (PFS) at 1 and 2 years from treatment initiation | 5 years
  Progression free survival will be measured as the length of time from treatment to progression of disease as measured by radiologic evaluation
To measure the duration of response (DOR) for the period of 2 years | 2 years
  DOR will be length of time from initial response to tumor progression documented by radiologic evaluation

OTHER OUTCOMES:
To evaluate the frequency of NPM/ALK quantitative polymerase chain reaction (qPCR) positivity in plasma | 2 years
  Detection of the NPM/ALK fusion gene via quantitative PCR (qPCR) in plasma
The evaluate the persistence of NPM/ALK DNA construct in plasma and correlation with rate of relapse | 2 years
  NPM-ALK DNA construct in plasma will be measured prospectively by polymerase chain reaction
To evaluate for ALK mutations in tumor and plasma at baseline and at time of relapse | 2 years
  ALK mutations in tumor and plasma will be analyzed by next generation sequencing
Changes in ALK-dependent NF-kB activation | 2 years
  NFKB1 and NFKB2 nuclear translocation/accumulation will be tested by immune histochemistry (IHC)
Changes in ALK phosphorylation | 2 years
  ALK phosphorylation (indicator of brigatinib efficacy) will be tested by immune histochemistry (IHC)
Changes in TRAF2 expression | 2 years
  TRAF2 expression (E3 ligase required for ALK mediation of NF-kB activation) will be tested by immune histochemistry (IHC)
To evaluate gene expression profiles before and after treatment with brigatinib | 2 years
  Gene expression profiling of NF-kB will be performed in tumor before and after treatment with brigatinib

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States